CLINICAL TRIAL: NCT04240860
Title: Randomized Clinical Trial Between Autologous Intrauterine Platelet-Rich Plasma Instillation And Three Snip Hysteroscopic Endometrial Scratching for Thinned Endometrium
Brief Title: Autologous Intrauterine Platelet-Rich Plasma Instillation And Endometrial Scratching for Thinned Endometrium
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed Mohsen Ahmed Mostafa Abo elnasr, resident in obs gyn department, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: prp thinned endometrium
Record Dates: First submitted 2019-09-13; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Infertility Due to Nonimplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich plasma preparation (Experimental): * About 15 ml of autologous blood from the patient was collected slowly in 20 ml syringe containing 1.5 ml anticoagulant citrate dextrose solution A (ACDA) under complete aseptic precautions.
    2- Blood was mixed by swinging the syringe slowly. 3- By using 18G needle, the gathered blood was transfused into tube maintaining a slope of 45°.
    4- The centrifugation step was then done by using non digital angle type centrifuge :the tube was put with water tube on the opposite side to achieve centrifuge balance.
    5- The centrifugation occurred in one step by power 3600 RPM for 6 minutes. 6- The buffy coat was elevated up to the buffy coat line (Figure 1). 7- the buffy coat (2-3 ml PRP) was extracted from slim neck by tornado technique so that sunk platelets can be floated and drawn easily.
    8- the remaining platelet poor plasma(PPP) was drawn using 5 cc syringe. then inserted by ovum pick up needle into subendometrium
  Interventions: Biological: platlet rich plasma
- endometrial scratch (Active Comparator): using scissor of hysteroscopr 3 snips was done in the fundus
  Interventions: Procedure: endometrial scratch

INTERVENTIONS:
Biological: platlet rich plasma — Drug: PRP PRP subendometrial infusion
  Device: ovum oickup needle PRP subendometrial infusion by hysteroscopic guided ovum pickup needle day 9 of the cycle
  Arms: platelet rich plasma preparation
Procedure: endometrial scratch — Three Snip Hysteroscopic Endometrial Scratching in luteal phase of preceeding cycle
  Arms: endometrial scratch

SUMMARY:
aim of that study is to compare the effect between autologous intrauterine Platelet-Rich Plasma instillation and three snip hysteroscopic endometrial scratching for thinned endometrium.

DETAILED DESCRIPTION:
Embryo implantation is a very delicate and well-orchestrated process that is governed by the interaction between several maternal and embryonic factors, ultimately resulting in adherence of the blastocyst to the endometrium. For a short period of time during the normal menstrual cycle, the endometrium represents the fertile "soil" for the implanting embryo. The human endometrium undergoes complex changes, in response to circulating estrogen and progesterone, which culminate at the mid-luteal phase of the menstrual cycle when it becomes suitable to host the blastocyst.

In clinical practice, a thin endometrium, unresponsive to conventional therapies, usually results in cycle cancellation and embryo cryopreservation. The evaluation of an adequate endometrial growth is performed using grey-scale ultrasound. The minimal endometrial thickness required for embryo transfer is now considered about 7 mm at the end of natural or medically induced follicular phase Local injury to the endometrium has been proposed as a means to improve implantation in women with RIF. Initial non-randomized studies showed a doubling of implantation rates after 2-4 endometrial injuries performed at different time points of the menstrual cycle in women with previous implantation failure . Following that, a number of randomized trials focusing on women with RIF have been conducted. The majority of the trials have demonstrated significant improvements in implantation rates, clinical pregnancy rates and/or live birth rates following endometrial injury performed in the preceding cycle Platelet rich plasma (PRP) represents a relatively new approach in regenerative medicine. It is obtained from patient's own blood and contains different growth factors and other biomolecules necessary for wound healing. Platelet rich plasma (PRP) therapy has accumulated considerable attention over the two last decades, mainly due to its potential ability in regenerative medicine. Platelets as a main components of the PRP, contain more than 1100 different proteins, with numerous post-translational modifications, resulting in over 1500 protein-based bioactive factors These factors include immune system messengers, growth factors, enzymes and their inhibitors and factors which can participate in tissue repair and wound healing. Another important characteristic of PRP is that represents an autologous product, which is prepared from the patient's own blood. Therefore, the use of autologous PRP eliminates any concerns about the risk of crossed contamination, disease transmission or immune reactions

ELIGIBILITY:
Inclusion Criteria:

Endometrial thickness < 7 mm under estrogen replacement therapy or repeated implantation failure Age between 18 and 38years

Exclusion Criteria:

Age < 18 and > 46 years Pregnancy Bleeding diathesis Previous uterine surgery (miomectomy, cesarean section, etc...) Platelet count < 105/μL Hemoglobin < 10 g/dL Presence of a tumor in the wound bed or metastatic disease Current diagnosis of cancer Other concomitant active infections Other factors of infertility ( PCO, tubal block, congenital anomalies, genetic malformation, male infertility)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 40 (Estimated)
Dates: Start 2020-01-23 (Estimated); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | 24-48h after intervention
  Endometrial thickness > 7 mm measured by means of transvaginal ultrasound

SECONDARY OUTCOMES:
Positive pregnancy test rate | Approximately 4 weeks after treatment
  Positive pregnancy test rate

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Farrag, Ph.D, Study Chair — professor; Elham H Madney, Ph.D, Study Director — assisted professor; Rasha E Khamiss, PH.D, Principal Investigator — lecturar

REFERENCES:
- [Background] Zadehmodarres S, Salehpour S, Saharkhiz N, Nazari L. Treatment of thin endometrium with autologous platelet-rich plasma: a pilot study. JBRA Assist Reprod. 2017 Feb 1;21(1):54-56. doi: 10.5935/1518-0557.20170013. PMID 28333034
- [Background] Molina A, Sanchez J, Sanchez W, Vielma V. Platelet-rich plasma as an adjuvant in the endometrial preparation of patients with refractory endometrium. JBRA Assist Reprod. 2018 Mar 1;22(1):42-48. doi: 10.5935/1518-0557.20180009. PMID 29303234
- [Background] Tandulwadkar SR, Naralkar MV, Surana AD, Selvakarthick M, Kharat AH. Autologous Intrauterine Platelet-Rich Plasma Instillation for Suboptimal Endometrium in Frozen Embryo Transfer Cycles: A Pilot Study. J Hum Reprod Sci. 2017 Jul-Sep;10(3):208-212. doi: 10.4103/jhrs.JHRS_28_17. PMID 29142450
- [Background] Nastri CO, Ferriani RA, Raine-Fenning N, Martins WP. Endometrial scratching performed in the non-transfer cycle and outcome of assisted reproduction: a randomized controlled trial. Ultrasound Obstet Gynecol. 2013 Oct;42(4):375-82. doi: 10.1002/uog.12539. Epub 2013 Sep 2. PMID 23754314
- [Background] Shokeir T, Ebrahim M, El-Mogy H. Hysteroscopic-guided local endometrial injury does not improve natural cycle pregnancy rate in women with unexplained infertility: Randomized controlled trial. J Obstet Gynaecol Res. 2016 Nov;42(11):1553-1557. doi: 10.1111/jog.13077. Epub 2016 Jul 1. PMID 27363928